CLINICAL TRIAL: NCT05572177
Title: Feasibility of MHealth Technology for Improving Self-Management and Adherence Among Asthmatic Adolescents
Brief Title: Feasibility of a Smartphone Application for Asthma Self-management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY000956; R34HL145442 (NIH)
Record Dates: First submitted 2022-07-25; First posted 2022-10-07 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Asthma Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Asthma SMART (Experimental): Subjects randomized to the intervention arm will be provided with the app to download to their personal iPhone or Android smartphone. Subjects will be asked to use the app every day for 6 months.
  Interventions: Device: Asthma SMART
- Standard of care (No Intervention): Subjects randomized to the standard-of-care arm will continue to receive regular care for their condition.

INTERVENTIONS:
Device: Asthma SMART — The intervention is a smartphone application to improve self-management of asthma designed to appeal to adolescents. The app integrates four components to facilitate asthma self-management: 1) self-monitoring of peak-flow and symptoms; 2) graphical health user interfaces with avatars, infographics, and rewards; 3) interactive educational materials; and 4) patient-provider interactions.
  Arms: Asthma SMART

SUMMARY:
The primary goal of this project is to determine the feasibility, acceptability, and adherence of a smartphone application for improving asthma self-management in a pilot randomized controlled trial (RCT). The app is specifically designed to appeal to adolescents. Adolescents with persistent asthma will be randomized to receive: 1) standard-of-care or 2) the self-management app in addition to standard-of-care. Feasibility will be assessed by the ability to recruit and retain subjects, technical barriers to implementation, and the appropriateness of the intervention among adolescents and providers. The acceptability of the intervention will be determined by appraising perceived usefulness, entertainment, and ease of use of the app. Adherence to usage of the app over a 6-month period will be assessed by examining the frequency of app usage and the features that were used, and the extent of data regarding self-management that was entered. A secondary objective is to obtain preliminary estimates of effectiveness of the app on clinical outcomes (ACT score, spirometry, CHSA-C, exacerbations, and medication adherence) relative to standard-of-care. It is hypothesized that the app will result in a high level of adherence and will be a feasible and acceptable intervention to improve self-management among adolescents with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 and less than 18 years at enrollment
* Established mild, moderate, or severe persistent asthma with a diagnosis verified by clinic physicians
* Speak English
* Not planning on moving out of the Tampa Bay area during the trial period
* Must have a suitable iPhone or Android device available to use with the app

Exclusion Criteria:

* Having mental or other development disorder that may make self-management of a chronic condition difficult
* Having other chronic lung disease or one or more of the following disorders including cystic fibrosis, neuromuscular disease, immunodeficiency or autoimmune disorders, blindness or severe vision impairment that may interfere with the ability to use the mobile app
* Having participated in the app development phase of the funded project

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate (number recruited per month) | 6 months
  The recruitment rate will be defined as the total number of participants recruited divided by the number of months of recruitment to determine the approximate number of participants recruited in a single site per month.
Retention rate (proportion that complete the 6-month trial) | 6 months
  The retention rate will be calculated as the number of participants that complete the 6 month follow-up exam divided by the total number of participants randomized in the study.
Technical feasibility (percentage of screened population) | 6 months
  The percentage of the screened population that has a suitable smartphone and data plan or wi-fi access in order to use the app.
Mean overall usability score obtained from the Health-ITUES | Assessed at the end of the 6 month trial
  The Health Information Technology Usability Evaluation Scale is a validated survey of usability of mobile health technology consisting of 20 questions each on a 5-point Likert scale with four subscale domains on impact, perceived usefulness, perceived ease of use, and user control. The total score is calculated as the average score across the domains with a value range from 1 to 5. Higher scores represent greater usability.
Average app usage per day | 6 months
  Sustainability of app usage will be defined as the number of days each participant interacted with the app at least once divided by the total number of days in the trial. Interaction is defined as performing any activity in the app.
Adherence to app reminders (proportion of app reminders) | 6 months
  Adherence to the app will be determined by examining the frequency of responses to app reminders. Adherence will be calculated as the number of activities completed in response to an app reminder divided by the total number of reminders received.

SECONDARY OUTCOMES:
Change in ACT score from baseline to the 6-month end point | Baseline and 6 month end-point
  The ACT test is a validated 5-question survey used to measure asthma control according to NHLBI guidelines. Total scores range from 5 to 25. Change will be calculated as the 6-month ACT score - baseline ACT score.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Alman, PhD, Principal Investigator — University of South Florida; Marisa Couluris, DO, Principal Investigator — University of South Florida; Paul Rosen, PhD, Principal Investigator — University of Utah
Locations (1):
- University of South Florida, Tampa, Florida, United States